CLINICAL TRIAL: NCT06735638
Title: Outside the Cage (OTC) Robotic Esophagectomy , Single Center Phase I Trial
Brief Title: Outside the Cage (OTC) Robotic Esophagectomy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Moishe Liberman, MD, PhD, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-12036
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Minimally invasive esophagectomy (MIE); Robotic-assisted surgery; Phase I clinical trial; Outside the Cage (OTC) technique; Robotic-assisted thoracic surgery (RATS); Enhanced recovery after surgery (ERAS); Non-intercostal approach
MeSH Terms: conditions — Esophageal Neoplasms; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Out of the Cage Minimally Invasive Esophagectomy (OTC MIE) (Experimental): Consented patients will undergo minimally invasive esophagectomy (MIE) using the Out of the Cage (OTC) robotic approach. This approach follows the standard procedural steps typically used in minimally invasive esophagectomy (e.g., laparoscopy and robotic-assisted thoracic surgery), with the primary difference being the incisions. Instead of intercostal incisions, the thoracic component of the procedure will be performed using 1 to 4 subcostal ports, tailored to the patient's anatomy and the case requirements.
  Interventions: Procedure: OTC MIE Esophagectomy

INTERVENTIONS:
Procedure: OTC MIE Esophagectomy — Consenting patients will undergo minimally invasive esophagectomy (MIE) using the Out of the Cage (OTC) robotic-assisted technique. The procedure will follow the exact standard steps of traditional VATS/RATS esophagectomy, except the thoracic ports will be placed in the subcostal plane. The number of ports (1-4) will be determined based on the patient and case characteristics.
  The Da Vinci Xi® surgical system will be used to perform the thoracic portion of the esophagectomy through subcostal ports using the standard technique. Once the procedure is completed, the robotic arms and ports will be removed from the chest, and figure-of-8 stitches with non-absorbable sutures will be placed to close the diaphragm at the port sites. A 24 Fr soft chest tube will be left in place, as per standard VATS/RATS esophagectomy protocols. Incisions will be closed in the standard manner.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and safety of a novel non-intercostal robotic approach for minimally invasive esophagectomy (OTC MIE) in the treatment of esophageal cancer. This study aims to determine whether OTC MIE reduces the risk of acute and chronic chest pain compared to traditional minimally invasive esophagectomy (MIE) and improves postoperative outcomes for patients. Participants will undergo either the OTC MIE procedure or a traditional MIE approach as part of their treatment for esophageal cancer. Postoperative outcomes, including chest pain and recovery metrics, will be closely monitored. Follow-up assessments will be conducted to evaluate the long-term safety and effectiveness of the novel approach. The investigators aim to recruit 31 patients.

DETAILED DESCRIPTION:
Esophageal cancer is the seventh most common cancer diagnosis worldwide, with approximately 604,000 new cases in 2022. Esophagectomy remains a cornerstone of esophageal cancer treatment, typically combined with perioperative chemoradiation for locally advanced disease. The procedure can be performed using various approaches, including open surgery and minimally invasive esophagectomy (MIE). MIE combines laparoscopy with thoracic techniques such as video-assisted thoracic surgery (VATS) or robotic-assisted surgery (RA), aiming to minimize trauma and improve both postoperative and long-term outcomes.

While VATS and RA have demonstrated reduced cardiopulmonary morbidity and mortality compared to open esophagectomy, both methods still involve intercostal incisions. These incisions can cause trauma to intercostal nerves and bundles, potentially leading to acute and chronic postoperative chest pain. The evolution of minimally invasive techniques in thoracic and lung surgery has focused on reducing the size and number of incisions to minimize surgical trauma. However, even with these advancements, intercostal instrumentation remains a source of significant postoperative complications.

Our group has developed a novel non-intercostal robotic approach for thoracic surgery called Outside the Cage (OTC) RATS. This technique was successfully implemented in over 60 lung resections, with the first published series showing promising outcomes, including feasibility, safety, and reduced postoperative pain. Additionally, results from a phase I clinical trial (NCT05832112) confirmed the safety and feasibility of this approach, with trends indicating faster recovery and less postoperative pain. Based on this experience, we recently performed the world's first OTC esophagectomy and have since refined the technique with successful outcomes, including no conversions to open surgery, transfusions, or major complications.

This study is a prospective pilot phase I trial designed to assess the feasibility and safety of OTC MIE in patients treated for esophageal cancer. Patients eligible for participation will include those already scheduled for MIE based on clinical indications such as tumor size, location, and individual characteristics. By avoiding intercostal instrumentation, we hypothesize that the OTC MIE approach will positively impact postoperative outcomes, enhancing recovery and reducing complications.

The primary objective of this study is to evaluate the feasibility of performing OTC MIE. The secondary objective is to systematically analyze the safety and postoperative recovery of patients undergoing this technique.

This trial is timely given our institution's extensive experience with both traditional MIE and OTC RATS. The results of this study could have significant implications for clinical practice by demonstrating the benefits of a non-intercostal approach for esophageal cancer surgery, potentially improving patient recovery and reducing the burden on healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

All patients with clinical stage I, II, or III esophageal cancer (cT1-3N0-2M0) scheduled to undergo minimally invasive esophagectomy (MIE) by VATS/RATS at the CHUM.

Exclusion Criteria:

* Age < 18 years old
* Inability to consent to the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | Through study completion, an average of 1 year
  Feasibility will be evaluated by completion of the procedure without conversion of the approach or technique. Any change in the treatment plan requiring the use of intercostal ports, conversion to conventional minimally invasive thoracic surgery through intercostal incisions, or conversion to open surgery
30-day mortality | 30 days after discharge
  Safety will be evaluated by 30-day mortality. Any dead occurring during the hospital stay or within 30 days after discharge will be registered.

SECONDARY OUTCOMES:
Length of stay | Through study completion, an average of 1 year
  Length of hospital stay
Operative time | Intraoperative
  Surgical operative time including robot positioning
Estimated blood loss | Intraoperative
  Registered by the OR nurse team
Postoperative pain | Through study completion, an average of 1 year
  Pain scores on a visual analog scale: Pain Rating Scale between 0 and 10 (0: better outcome and 10:Worse outcome)
Quality of recovery | Through study completion, an average of 1 year
  Assessment of postoperative recovery using Quality Of Recovery (QOR-15) questionnaire between 0 and 10 (0: Better outcome and 10: Worst outcome)
Analgesic complementation requirement | Through study completion, an average of 1 year
  Number of participants who need of adding analgesia medication out of the analgesic pathway used in our center for conventional RATS/VATS
Serious adverse events | Through study completion, an average of 1 year
  Complications derived from the operation that altered the pathway
Perioperative complications | Through study completion, an average of 1 year
  Complications including intraoperative and postoperative occurring during the hospital stay or within 30 days after discharge will be graded according to the Clavien-Dindo classification
Evaluate Chronic Pain | Through study completion, an average of 1 year
  Pain scores on a visual analog scale: Pain Rating Scale between 0 and 10 (0: better outcome and 10:Worse outcome).
  Chronic pain of OTC RATS lobectomy patients will be compared to that of VATS lobectomy patients, for which the data will also be collected and analysed retrospectively.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No